CLINICAL TRIAL: NCT01347229
Title: Assessment of Sitting and Supine Position IOP Using SENSIMED Triggerfish® and Standard Tonometers
Brief Title: SENSIMED Triggerfish® in Sitting and Supine Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sensimed AG (Industry)
Responsible Party: Jeam-Marc Wismer, Sensimed AG
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10/06
Record Dates: First submitted 2011-05-02; First posted 2011-05-04 (Estimated); Last update posted 2012-04-17 (Estimated); Status verified 2012-04

CONDITIONS: Healthy Subjects
Keywords: Glaucoma; Triggerfish; body position
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: SENSIMED Triggerfish® — Soft contact lens-based device for the continuous monitoring of IOP fluctuations

SUMMARY:
The purpose of the study is to evaluate changes in intraocular pressure (IOP) between sitting and supine body positions and correlate the values obtained with conventional tonometers to the output provided by the investigational device.

DETAILED DESCRIPTION:
20 subjects will be enrolled in the investigation. Eligible subjects will receive one session of 22-hour continuous IOP monitoring with SENSIMED Triggerfish® in ambulatory mode, with body position transitions carried out in-hospital. SENSIMED Triggerfish® will be installed randomly on right or left eyes and the IOP recording will be initiated as soon as the adaptation of the device on the subject's eye is satisfying. Subjects will then go home. The next morning, subjects will return to the hospital and during SENSIMED Triggerfish® monitoring on one eye, IOP measurements will be taken in the fellow eye in sitting position using Goldmann, tonopen and pneuma-tonometers. Then subjects will lie down on a flat bed. After 15 ± 5 minutes and again after 45 ± 5 minutes IOP will be measured in supine position, using Goldmann, tonopen, pneuma-tonometer and Perkins tonometers. Then subjects will sit up again. After 30 ± 5 minutes IOP will be measured with the Goldmann tonometer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to provide informed consent
* Healthy subject, with no previous ocular medical history, with the exception of spectacle vision correction for myopia, hyperopia and astigmatism
* No more than 4 diopters spherical equivalent
* No more than 2 diopters cylinder equivalent
* GAT IOP of less than or equal to 21 mmHg at inclusion and open iridocorneal angles, no history of any IOP > 21 mmHg
* GAT IOP difference between eyes within 1 mmHg during initial exam
* GAT IOP differences between initial sitting and supine positions, between left and right eyes, within 2 mmHg during initial exam
* ≥ 18 years
* For women with childbearing potential, adequate contraception

Exclusion Criteria:

* Subjects with contraindications for wearing contact lenses
* Severe dry eye syndrome
* Keratoconus or other corneal abnormality
* Conjunctival or intraocular inflammation
* History of eye surgery
* Full frame metal glasses during SENSIMED Triggerfish® recording
* Known hypersensitivity to silicone, plaster or ocular anesthesia
* Pregnancy and lactation
* Simultaneous participation in other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-04; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference in study device signal and GAT IOP between the sitting and supine positions during the sitting-supine sequence | 45 minutes

SECONDARY OUTCOMES:
Difference in Triggerfish® signal and GAT IOP between the sitting and supine positions upon returning to sitting position from supine | 30 minutes
IOP measurements with tonopen and pneuma-tonometer in sitting position, and tonopen, pneuma-tonometer and Perkins in supine position | 2 hours
Monitoring with study device obtained before Day 2 | 20 hours

CONTACTS AND LOCATIONS:
Overall Officials: Yaniv Barkana, MD, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Assaf Harofeh Medical Center, Ẕerifin, Israel